CLINICAL TRIAL: NCT03278314
Title: Tezacaftor/Ivacaftor Combination Therapy Expanded Access Program for Patients 12 Years of Age and Older With Cystic Fibrosis
Status: Approved for marketing | Type: Expanded Access
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: VX17-661-901
Record Dates: First submitted 2017-09-06; First posted 2017-09-11 (Actual); Last update posted 2018-11-02 (Actual); Status verified 2018-10

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — tezacaftor, ivacaftor drug combination

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: tezacaftor/ivacaftor — orally administered TEZ/IVA combination therapy
  Other Names: TEZ/IVA

SUMMARY:
To provide TEZ/IVA combination therapy to CF patients who are 12 years of age and older who completed Vertex TEZ/IVA combination therapy clinical studies (NCT02565914 or NCT03150719). To provide TEZ/IVA combination therapy to CF patients in critical need who are 12 years of age and older, homozygous for F508del.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 12 years of age and older with confirmed diagnosis of CF.

  1. - completed Vertex clinical studies NCT02565914 or NCT03150719, or
  2. - are homozygous for F508del and have (1) discontinued Orkambi within 12 weeks from start of treatment because of the onset of respiratory AEs considered to be treatment related or (2) cannot initiate Orkambi because of chronic treatment with an essential sensitive CYP3A substrate or a CYP3A substrate with a narrow therapeutic index AND who meet at least 1 of the following criteria:

     * the highest percent predicted forced expiratory volume in 1 second (ppFEV1) is <40 in the 6 months before the date of completion of the request form, or
     * documentation of being active on a lung transplant waiting list or documentation of being evaluated for lung transplantation, but deemed unsuitable because of contraindications, or
     * rapid and persistent loss of lung function, defined as at least a 20% relative decrease in ppFEV1 in the last 6 months and sustained for at least 1 month despite appropriate treatment.

Exclusion Criteria:

* History of any comorbidity that, in the opinion of the treating physician, might pose undue risk in administering TEZ/IVA combination therapy to the patient (e.g., history of advanced liver disease).
* Ongoing or prior participation in an investigational drug study (with the exception of Vertex clinical studies evaluating TEZ/IVA) within 5 terminal half-lives of the previous investigational study drug or 30 days, whichever is longer, of first administration of TEZ/IVA.
* Subjects who are pregnant.
* Patients eligible for participation in ongoing clinical studies evaluating TEZ/IVA or other CFTR modulator therapies.

Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 12 Years | Sex: All
Age Groups: Child, Adult, Older Adult